CLINICAL TRIAL: NCT00891332
Title: Phase II Study of S-1 Plus LV (1 Week on and 1 Week Off) as First-line Treatment for Patients With Metastatic Colorectal Cancer
Brief Title: Study of S-1 Plus LV for Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Taiho10020400
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): S-1 plus LV
  Interventions: Drug: S-1 plus LV (The combination therapy of S-1 and Leucovorin)

INTERVENTIONS:
Drug: S-1 plus LV (The combination therapy of S-1 and Leucovorin) — S-1 40-60 mg bid day 1～day 7 LV 25 mg bid day 1～day 7

SUMMARY:
This is a multicenter study designed to evaluate the response rate of S-1 plus Leucovorin (1 week on and 1 week off) as first -line treatment for patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved adenocarcinoma
* Unresectable and recurrent colorectal cancer
* Age20 ≤ at enrollment
* Performance status 0 or 1 (ECOG)
* No prior treatment (ex. radiation therapy, chemotherapy, hormonal therapy) to advanced disease. Patients who received adjuvant chemotherapy more than 180 days before enrollment can be allowed but those who received S-1 containing treatment shall be excluded
* Adequate hematologic, hepatic and renal functions
* At least one measurable lesion by RECIST criteria

Exclusion Criteria:

* Serious drug hypersensitivity
* Pregnant or nursing
* Bleeding from gastrointestinal tract
* Diarrhea
* Simultaneously active double cancer
* Serious illness or medical condition
* Brain metastasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | During chemotherapy

SECONDARY OUTCOMES:
Safety | During chemotherapy
Progression free survival (PFS) | Until progression
Disease control rate(DCR) | During chemotherapy
Time to treatment failure (TTF) | Until progression
Overall survival (OS) | Over two years from registration
Feasibility | During chemotherapy
Pharmacokinetics | During chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hideo Baba, M.D., Principal Investigator — Graduate School of Medical Sciences Kumamoto University
Locations (6):
- China (5):
  - Sun Yat-sen University Cancer Center, Division of Oncology, Dong Feng Dong road,Guangzhou, Guangdong
  - Shanghai Fudan University Cancer Hospital, Division of Oncology, Dong An Road, Shanghai
  - PLA 307 Hospital, No.4 Division of Oncology, East Avenue, Fengtai District, Beijing
  - Beijing Cancer Hospital, Digestive System Medicine Department, Fucheng Road, Haidian District, Beijing
  - Cancer Institute & Hospital Chinese Academy of Medical Sciences, Division of Oncology, Panjiayuan Nanli, Chaoyang District, Beijing
- Graduate School of Medical Sciences Kumamoto University, 1-1-1, Honjo Kumamoto-city, Kumamoto, Japan